CLINICAL TRIAL: NCT05385289
Title: A Cognitive-behavioral Approach of Rumination as Intervention for Overgeneral Mode of Processing in Perfectionism: a Single-case Experimental Design
Brief Title: A Cognitive-behavioral Intervention of Rumination for Perfectionists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/17JAN/016
Record Dates: First submitted 2022-03-24; First posted 2022-05-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Perfectionism; Rumination - Thoughts; Anxiety; Depression
Keywords: Perfectionism; Rumination; Autobiographical Memory; Overgeneral processing; SCED
MeSH Terms: conditions — Anxiety Disorders; Depression; Rumination Syndrome | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The final sample will comprise 12 participants.
  The initial sample size was based on Shadish & Sullivan's (2011) study reporting that the median and modal number of participants in single-case designs is three. Therefore, recruiting 6 participants allowed for a direct intrasubject replication (i.e., a "replication of the experimental effect within the design") while ensuring that three participants were retained despite possible dropout. Moreover, using two waves of six participants (resulting in a total sample of 12 participants) allowed for a direct inter-subject replication (i.e., "repeating the same study but with additional individuals"). Those two replications were used to demonstrate that changes on target behaviors systematically arrives after the intervention introduction, hence controlling for external variables.
Masking Description: A computerized version of the Autobiographical Memory Test (AMT; Williams et Broadbent, 1986) will be used to assess the overgeneral processing. This task focused on retrieving past memories of personal events.
  AMT raters will be not involved in any other aspect of the study procedures. The memories will also be presented to the raters in a randomized order, so that there was no possibility of guessing who completed them or when.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First wave with 6 participants (Experimental): Once selected, an individual online information session will be scheduled with each selected participant to explain the project and its practical implications. At this time, six of the twelve participants will be provided a link to complete online measures as the A-baseline phase, to constitute their own non-intervention control condition on the target behavior (i.e., rumination) and on positive and negative emotions. The other six participants will be entered into a 3-week waiting list period with a sequential introduction, to provide another non-intervention control condition.
  The A-baseline phase length will include at least 5 measures and most 10 measures, resulting in 10 potential starting point for the B-experimental phase. This range will be determined to estimate autocorrelation and its associated bias.
  Interventions: Behavioral: A cognitive-behavioral approach of rumination as intervention for overgeneral mode of processing in perfectionism
- Second wave with 6 other participants (Experimental): After three weeks, the six participants on the waiting list will also begin the same A-baseline phase as the six participants of the first wave.
  Interventions: Behavioral: A cognitive-behavioral approach of rumination as intervention for overgeneral mode of processing in perfectionism

INTERVENTIONS:
Behavioral: A cognitive-behavioral approach of rumination as intervention for overgeneral mode of processing in perfectionism — The B-experimental phase consists in a 6-session intervention targeting rumination and lasting for 3 weeks. The intervention was derived from 3 manuals: Rumination-Focused Cognitive-Behavioral Therapy for Depression (Watkins, 2016), Overcoming Perfectionism (Shafran et al., 2010), and Cognitive-Behavioral Treatment of Perfectionism (Egan et al., 2014). Participants will attend 2 sessions per week at home. Each week will end with an individual 30 minutes-debriefing session with an experimenter, to ascertain understanding of session content and homework.
  Intervention sessions will be given in paper format to participant after the A-baseline-phase. A paper diary was also provided for homework, in addition to the session content caneva. Each session contains (a) theoretical content on ruminations linked to perfectionism, (b) exercises to create alternative habits to ruminations, and (c) homework to become aware of ruminations and to experiment with alternatives.

SUMMARY:
This study aims to investigate the mediating role of rumination in the relationship between perfectionism and psychological distress, by proposing a cognitive-behavioral intervention targeting rumination. This intervention aims at decreasing - or even neutralizing - the effect of the mediator and then examining how this decrease impacts the relationship between perfectionism and psychological distress.

A randomized, concurrent, multiple-baseline single-case design will be applied.

DETAILED DESCRIPTION:
Perfectionism is defined as "exceedingly high standards of performance accompanied by critical evaluations of oneself and others and a fear of negative social evaluation if not perfect". Factorial analyses of the two main perfectionism scales have identified two overarching dimensions: Perfectionistic Strivings and Perfectionistic Concerns. The perfectionistic concerns dimension is generally associated with negative outcomes and psychopathology, while perfectionistic strivings have been found to yield both positive outcomes and negative outcomes.

Perfectionism is a central transdiagnostic phenomenon involved in the maintenance of multiple psychological disorders (e.g., anorexia nervosa, obsessive compulsive disorder, chronic fatigue, and depression). After decades of research focusing on scales development or relying exclusively on correlational studies, the experimental investigation of the processes underlying perfectionism is just emerging. On a theoretical basis, two processes related to emotional information processing seem particularly relevant: rumination and autobiographical memory. The objective of this study is to investigate with a randomized, concurrent, multiple-baseline single-case design the contribution of these processes to perfectionists' psychological vulnerability.

Rumination is defined as a mental process characterized by repetitive, prolonged, and recurrent thinking about one's concerns and one's experience. The control theory suggests that individuals engage in rumination when perceiving a discrepancy between their goals and their current condition, and stay in this mode of thinking until the goal is either attained or abandoned. Based on this theoretical background, recent research suggests that rumination could be one of the processes explaining the perfectionistic vulnerability to psychological distress, by perseveringly focusing on the discrepancy between high and demanding standards and the actual performance. However, only few study has experimentally manipulated this process, thus precluding from any causal inference.

Autobiographical memories are "memories about personal experiences that go beyond the mere factual description of the event to include personal beliefs, emotions, and thoughts". One feature of those memories is the specificity level defined as "the extent to which retrieved autobiographical memories are specific or not (i.e., memory of a particular event that happened at a particular time and place that lasted no more than one day). Difficulty with retrieving such specific memories is called overgeneral autobiographical memory".

The perfectionism cognition theory aims to clarify how autobiographical memory and working memory might be affected by perfectionist tendencies. It especially postulates retroactive loops between (a) repetitive thinking, (b) an overdeveloped memory for mistakes, failures, and stressful experiences, and (c) a hypervigilance and cognitive bias toward related cues that signal the possibility of failure, mistakes, and negative social evaluation. These authors suggested that perfectionists are characterized by deficits in attentional capacity and working memory during times of stress. This promising cognitive approach has partially been supported. For example, a recent meta-analysis states that perseverative cognitions (i.e., worry and rumination) mediate the relationship between perfectionism and distress in non-clinical samples. However, empirical evidence of an experimental nature is still needed, in particular for the postulated autobiographical memory and working memory biases.

To overcome those limitations, the present study will manipulate rumination with a clinical intervention, to block its mediational role on the relationship between perfectionism and psychological distress (here operationalized by mood state and anxio-depressive symptoms). Moreover, this study aims to go further than identifying a true mediator: its aims to explain the mechanism "through which change come about", namely through a concreteness training to overcome overgeneral mode of processing. Indeed, even if the main focus of the study is to identify mediators that may statistically account for the relationship between perfectionism and psychological distress, a ideal purpose is to propose a therapeutic intervention that may target mechanisms of change underlying hypothesized mediator.

ELIGIBILITY:
Inclusion Criteria:

* Being native French speakers
* Reporting significant levels of (1) perfectionism, (2) abstract and evaluative repetitive thinking, and (3) anxio-depressive symptoms.

Exclusion Criteria:

* Being involved in a therapeutic treatment.
* Being under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Perfectionism - Hewitt and Flett's Multidimensional Perfectionism Scale (HMPS; Hewitt & Flett,1991) | For the recruitment, i.e. until the number of 6 participants is reached for the second wave of the study (approximately two months after the beginning of the study)
  The HMPS includes 45 items assessing the three following subdimensions: Self-Oriented Perfectionism (SOP, reflecting "setting exacting standards for oneself and stringently evaluating and censuring one's own behavior" in the present study), Socially Prescribed Perfectionism (SPP, reflecting "the perceived need to attain standards and expectations prescribed by significant others"), and Other-Oriented Perfectionism (OOP, reflecting "unrealistic standards for significant others, places importance on other people being perfect, and stringently evaluates others' performance"). Participants completed the questionnaire with a Likert type scale ranging from 1 ("totally disagree") to 7 ("totally agree").
Perfectionism - Hewitt and Flett's Multidimensional Perfectionism Scale (HMPS; Hewitt & Flett,1991) | The day before the beginning of the intervention
  The HMPS includes 45 items assessing the three following subdimensions: Self-Oriented Perfectionism (SOP, reflecting "setting exacting standards for oneself and stringently evaluating and censuring one's own behavior" in the present study), Socially Prescribed Perfectionism (SPP, reflecting "the perceived need to attain standards and expectations prescribed by significant others"), and Other-Oriented Perfectionism (OOP, reflecting "unrealistic standards for significant others, places importance on other people being perfect, and stringently evaluates others' performance"). Participants completed the questionnaire with a Likert type scale ranging from 1 ("totally disagree") to 7 ("totally agree").
Perfectionism - Hewitt and Flett's Multidimensional Perfectionism Scale (HMPS; Hewitt & Flett,1991) | Once participants have completed 4 sessions of the intervention, about a week and a half after the beginning of the intervention
  The HMPS includes 45 items assessing the three following subdimensions: Self-Oriented Perfectionism (SOP, reflecting "setting exacting standards for oneself and stringently evaluating and censuring one's own behavior" in the present study), Socially Prescribed Perfectionism (SPP, reflecting "the perceived need to attain standards and expectations prescribed by significant others"), and Other-Oriented Perfectionism (OOP, reflecting "unrealistic standards for significant others, places importance on other people being perfect, and stringently evaluates others' performance"). Participants completed the questionnaire with a Likert type scale ranging from 1 ("totally disagree") to 7 ("totally agree").
Perfectionism - Hewitt and Flett's Multidimensional Perfectionism Scale (HMPS; Hewitt & Flett,1991) | Two weeks after the end of the intervention
  The HMPS includes 45 items assessing the three following subdimensions: Self-Oriented Perfectionism (SOP, reflecting "setting exacting standards for oneself and stringently evaluating and censuring one's own behavior" in the present study), Socially Prescribed Perfectionism (SPP, reflecting "the perceived need to attain standards and expectations prescribed by significant others"), and Other-Oriented Perfectionism (OOP, reflecting "unrealistic standards for significant others, places importance on other people being perfect, and stringently evaluates others' performance"). Participants completed the questionnaire with a Likert type scale ranging from 1 ("totally disagree") to 7 ("totally agree").
Perfectionism - Hewitt and Flett's Multidimensional Perfectionism Scale (HMPS; Hewitt & Flett,1991) | Three months after the end of the intervention
  The HMPS includes 45 items assessing the three following subdimensions: Self-Oriented Perfectionism (SOP, reflecting "setting exacting standards for oneself and stringently evaluating and censuring one's own behavior" in the present study), Socially Prescribed Perfectionism (SPP, reflecting "the perceived need to attain standards and expectations prescribed by significant others"), and Other-Oriented Perfectionism (OOP, reflecting "unrealistic standards for significant others, places importance on other people being perfect, and stringently evaluates others' performance"). Participants completed the questionnaire with a Likert type scale ranging from 1 ("totally disagree") to 7 ("totally agree").
Perfectionism - Frost, Marten, Lahart, and Rosenblate's Multidimensional Perfectionism Scale (FMPS; Frost, Marten, Lahart, and Rosenblate, 1990) | For the recruitment, i.e. until the number of 6 participants is reached for the second wave of the study (approximately two months after the beginning of the study)
  The FMPS is a 35-item questionnaire assessing six subdimensions: Concern Over Mistakes (CM, reflecting "negative reactions to mistakes, a tendency to interpret mistakes as equivalent to failure, and a tendency to believe that one will lose the respect of others following failure"), Personal Standards (PS, reflecting "the setting of very high standards and the excessive importance placed on these high standards for self-evaluation"), Doubts About Actions (DA, reflecting "the tendency to feel that projects are not completed to satisfaction"), Parental Expectations (PE, reflecting "the tendency to believe that one's parents set very high goals and are overly critical"), Parental Criticism (PC, reflecting "the perception of high parental criticism"), and Organization (O, reflecting "the emphasis on the importance of and preference for order and organization"). Participants completed the questionnaire with a Likert type scale ranging from 1 ("strongly disagree") to 5 ("strongly agree").
Perfectionism - Frost, Marten, Lahart, and Rosenblate's Multidimensional Perfectionism Scale (FMPS; Frost, Marten, Lahart, and Rosenblate, 1990) | The day before the beginning of the intervention
  The FMPS is a 35-item questionnaire assessing six subdimensions: Concern Over Mistakes (CM, reflecting "negative reactions to mistakes, a tendency to interpret mistakes as equivalent to failure, and a tendency to believe that one will lose the respect of others following failure"), Personal Standards (PS, reflecting "the setting of very high standards and the excessive importance placed on these high standards for self-evaluation"), Doubts About Actions (DA, reflecting "the tendency to feel that projects are not completed to satisfaction"), Parental Expectations (PE, reflecting "the tendency to believe that one's parents set very high goals and are overly critical"), Parental Criticism (PC, reflecting "the perception of high parental criticism"), and Organization (O, reflecting "the emphasis on the importance of and preference for order and organization"). Participants completed the questionnaire with a Likert type scale ranging from 1 ("strongly disagree") to 5 ("strongly agree").
Perfectionism - Frost, Marten, Lahart, and Rosenblate's Multidimensional Perfectionism Scale (FMPS; Frost, Marten, Lahart, and Rosenblate, 1990) | Once participants have completed 4 sessions of the intervention, about a week and a half after the beginning of the intervention
  The FMPS is a 35-item questionnaire assessing six subdimensions: Concern Over Mistakes (CM, reflecting "negative reactions to mistakes, a tendency to interpret mistakes as equivalent to failure, and a tendency to believe that one will lose the respect of others following failure"), Personal Standards (PS, reflecting "the setting of very high standards and the excessive importance placed on these high standards for self-evaluation"), Doubts About Actions (DA, reflecting "the tendency to feel that projects are not completed to satisfaction"), Parental Expectations (PE, reflecting "the tendency to believe that one's parents set very high goals and are overly critical"), Parental Criticism (PC, reflecting "the perception of high parental criticism"), and Organization (O, reflecting "the emphasis on the importance of and preference for order and organization"). Participants completed the questionnaire with a Likert type scale ranging from 1 ("strongly disagree") to 5 ("strongly agree").
Perfectionism - Frost, Marten, Lahart, and Rosenblate's Multidimensional Perfectionism Scale (FMPS; Frost, Marten, Lahart, and Rosenblate, 1990) | Two weeks after the end of the intervention
  The FMPS is a 35-item questionnaire assessing six subdimensions: Concern Over Mistakes (CM, reflecting "negative reactions to mistakes, a tendency to interpret mistakes as equivalent to failure, and a tendency to believe that one will lose the respect of others following failure"), Personal Standards (PS, reflecting "the setting of very high standards and the excessive importance placed on these high standards for self-evaluation"), Doubts About Actions (DA, reflecting "the tendency to feel that projects are not completed to satisfaction"), Parental Expectations (PE, reflecting "the tendency to believe that one's parents set very high goals and are overly critical"), Parental Criticism (PC, reflecting "the perception of high parental criticism"), and Organization (O, reflecting "the emphasis on the importance of and preference for order and organization"). Participants completed the questionnaire with a Likert type scale ranging from 1 ("strongly disagree") to 5 ("strongly agree").
Perfectionism - Frost, Marten, Lahart, and Rosenblate's Multidimensional Perfectionism Scale (FMPS; Frost, Marten, Lahart, and Rosenblate, 1990) | Three months after the end of the intervention
  The FMPS is a 35-item questionnaire assessing six subdimensions: Concern Over Mistakes (CM, reflecting "negative reactions to mistakes, a tendency to interpret mistakes as equivalent to failure, and a tendency to believe that one will lose the respect of others following failure"), Personal Standards (PS, reflecting "the setting of very high standards and the excessive importance placed on these high standards for self-evaluation"), Doubts About Actions (DA, reflecting "the tendency to feel that projects are not completed to satisfaction"), Parental Expectations (PE, reflecting "the tendency to believe that one's parents set very high goals and are overly critical"), Parental Criticism (PC, reflecting "the perception of high parental criticism"), and Organization (O, reflecting "the emphasis on the importance of and preference for order and organization"). Participants completed the questionnaire with a Likert type scale ranging from 1 ("strongly disagree") to 5 ("strongly agree").
Depression - Center for Epidemiologic Studies - Depression (CES-D; Radloff, 1997) | For the recruitment, i.e. until the number of 6 participants is reached for the second wave of the study (approximately two months after the beginning of the study)
  The CES-D is a 20-item questionnaire with a Likert type scale ranging to 0 ["rarely or none of the time (less than 1 day)"] to 3 ["most or all of the time (5-7 days)"]. It assesses the frequency of the main symptoms of depression over the past week. Those symptoms are categorized into four subscales: depressed affect (DA), positive affect (PA), somatic complaints (SC), and disturbed interpersonal relationships (IR).
Depression - Center for Epidemiologic Studies - Depression (CES-D; Radloff, 1997) | The day before the beginning of the intervention
  The CES-D is a 20-item questionnaire with a Likert type scale ranging to 0 ["rarely or none of the time (less than 1 day)"] to 3 ["most or all of the time (5-7 days)"]. It assesses the frequency of the main symptoms of depression over the past week. Those symptoms are categorized into four subscales: depressed affect (DA), positive affect (PA), somatic complaints (SC), and disturbed interpersonal relationships (IR).
Depression - Center for Epidemiologic Studies - Depression (CES-D; Radloff, 1997) | Once participants have completed 4 sessions of the intervention, about a week and a half after the beginning of the intervention
  The CES-D is a 20-item questionnaire with a Likert type scale ranging to 0 ["rarely or none of the time (less than 1 day)"] to 3 ["most or all of the time (5-7 days)"]. It assesses the frequency of the main symptoms of depression over the past week. Those symptoms are categorized into four subscales: depressed affect (DA), positive affect (PA), somatic complaints (SC), and disturbed interpersonal relationships (IR).
Depression - Center for Epidemiologic Studies - Depression (CES-D; Radloff, 1997) | Two weeks after the end of the intervention
  The CES-D is a 20-item questionnaire with a Likert type scale ranging to 0 ["rarely or none of the time (less than 1 day)"] to 3 ["most or all of the time (5-7 days)"]. It assesses the frequency of the main symptoms of depression over the past week. Those symptoms are categorized into four subscales: depressed affect (DA), positive affect (PA), somatic complaints (SC), and disturbed interpersonal relationships (IR).
Depression - Center for Epidemiologic Studies - Depression (CES-D; Radloff, 1997) | Three months after the end of the intervention
  The CES-D is a 20-item questionnaire with a Likert type scale ranging to 0 ["rarely or none of the time (less than 1 day)"] to 3 ["most or all of the time (5-7 days)"]. It assesses the frequency of the main symptoms of depression over the past week. Those symptoms are categorized into four subscales: depressed affect (DA), positive affect (PA), somatic complaints (SC), and disturbed interpersonal relationships (IR).
Anxiety - Generalized Anxiety Disorder Screener (GAD-7; Spitzer, Kroenke, Williams, Löwe, 2008) | For the recruitment, i.e. until the number of 6 participants is reached for the second wave of the study (approximately two months after the beginning of the study)
  The GAD-7 is a seven-items questionnaire with a Likert type scale ranging from 0 ("not at all") to 3 ("nearly every day"). It assesses the presence and the severity of the Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) symptom criteria for Generalized Anxiety Disorder over the past week.
Anxiety - Generalized Anxiety Disorder Screener (GAD-7; Spitzer, Kroenke, Williams, Löwe, 2008) | The day before the beginning of the intervention
  The GAD-7 is a seven-items questionnaire with a Likert type scale ranging from 0 ("not at all") to 3 ("nearly every day"). It assesses the presence and the severity of the Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) symptom criteria for Generalized Anxiety Disorder over the past week.
Anxiety - Generalized Anxiety Disorder Screener (GAD-7; Spitzer, Kroenke, Williams, Löwe, 2008) | Once participants have completed 4 sessions of the intervention, about a week and a half after the beginning of the intervention
  The GAD-7 is a seven-items questionnaire with a Likert type scale ranging from 0 ("not at all") to 3 ("nearly every day"). It assesses the presence and the severity of the Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) symptom criteria for Generalized Anxiety Disorder over the past week.
Anxiety - Generalized Anxiety Disorder Screener (GAD-7; Spitzer, Kroenke, Williams, Löwe, 2008) | Two weeks after the end of the intervention
  The GAD-7 is a seven-items questionnaire with a Likert type scale ranging from 0 ("not at all") to 3 ("nearly every day"). It assesses the presence and the severity of the Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) symptom criteria for Generalized Anxiety Disorder over the past week.
Anxiety - Generalized Anxiety Disorder Screener (GAD-7; Spitzer, Kroenke, Williams, Löwe, 2008) | Three months after the end of the intervention
  The GAD-7 is a seven-items questionnaire with a Likert type scale ranging from 0 ("not at all") to 3 ("nearly every day"). It assesses the presence and the severity of the Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) symptom criteria for Generalized Anxiety Disorder over the past week.
Rumination trait - Repetitive Thinking Mode Questionnaire (RTMQ; Philippot, Verschuren, & Douilliez, in press). | For the recruitment, i.e. until the number of 6 participants is reached for the second wave of the study (approximately two months after the beginning of the study)
  The RTMQ is a 18-item questionnaire, with a Likert type scale ranging from 1 ("almost never") to 4 ("almost always"). It assesses three dimensions of repetitive thinking processes : (a) abstract evaluative mode of repetitive thinking (AERT; " thoughts at an abstract, overgeneral level that address the causes and consequence of one's mood or condition, oriented toward the past and future rather than toward the present moment"), (b) concrete experiential mode of repetitive thinking (CERT; " mode of thinking centered on how one is presently feeling and experiencing the ongoing situation, and how a present experience unfolds"), and (c) creative dendritic mode of repetitive thinking (CDRT; "extremely fluent and flexible thinking, with creative content [new and original ideas], not necessarily centered on here and now experience".
Rumination trait - Repetitive Thinking Mode Questionnaire (RTMQ; Philippot, Verschuren, & Douilliez, in press). | The day before the beginning of the intervention
  The RTMQ is a 18-item questionnaire, with a Likert type scale ranging from 1 ("almost never") to 4 ("almost always"). It assesses three dimensions of repetitive thinking processes : (a) abstract evaluative mode of repetitive thinking (AERT; " thoughts at an abstract, overgeneral level that address the causes and consequence of one's mood or condition, oriented toward the past and future rather than toward the present moment"), (b) concrete experiential mode of repetitive thinking (CERT; " mode of thinking centered on how one is presently feeling and experiencing the ongoing situation, and how a present experience unfolds"), and (c) creative dendritic mode of repetitive thinking (CDRT; "extremely fluent and flexible thinking, with creative content [new and original ideas], not necessarily centered on here and now experience".
Rumination trait - Repetitive Thinking Mode Questionnaire (RTMQ; Philippot, Verschuren, & Douilliez, in press). | Once participants have completed 4 sessions of the intervention, about a week and a half after the beginning of the intervention
  The RTMQ is a 18-item questionnaire, with a Likert type scale ranging from 1 ("almost never") to 4 ("almost always"). It assesses three dimensions of repetitive thinking processes : (a) abstract evaluative mode of repetitive thinking (AERT; " thoughts at an abstract, overgeneral level that address the causes and consequence of one's mood or condition, oriented toward the past and future rather than toward the present moment"), (b) concrete experiential mode of repetitive thinking (CERT; " mode of thinking centered on how one is presently feeling and experiencing the ongoing situation, and how a present experience unfolds"), and (c) creative dendritic mode of repetitive thinking (CDRT; "extremely fluent and flexible thinking, with creative content [new and original ideas], not necessarily centered on here and now experience".
Rumination trait - Repetitive Thinking Mode Questionnaire (RTMQ; Philippot, Verschuren, & Douilliez, in press). | Two weeks after the end of the intervention
  The RTMQ is a 18-item questionnaire, with a Likert type scale ranging from 1 ("almost never") to 4 ("almost always"). It assesses three dimensions of repetitive thinking processes : (a) abstract evaluative mode of repetitive thinking (AERT; " thoughts at an abstract, overgeneral level that address the causes and consequence of one's mood or condition, oriented toward the past and future rather than toward the present moment"), (b) concrete experiential mode of repetitive thinking (CERT; " mode of thinking centered on how one is presently feeling and experiencing the ongoing situation, and how a present experience unfolds"), and (c) creative dendritic mode of repetitive thinking (CDRT; "extremely fluent and flexible thinking, with creative content [new and original ideas], not necessarily centered on here and now experience".
Rumination trait - Repetitive Thinking Mode Questionnaire (RTMQ; Philippot, Verschuren, & Douilliez, in press). | Three months after the end of the intervention
  The RTMQ is a 18-item questionnaire, with a Likert type scale ranging from 1 ("almost never") to 4 ("almost always"). It assesses three dimensions of repetitive thinking processes : (a) abstract evaluative mode of repetitive thinking (AERT; " thoughts at an abstract, overgeneral level that address the causes and consequence of one's mood or condition, oriented toward the past and future rather than toward the present moment"), (b) concrete experiential mode of repetitive thinking (CERT; " mode of thinking centered on how one is presently feeling and experiencing the ongoing situation, and how a present experience unfolds"), and (c) creative dendritic mode of repetitive thinking (CDRT; "extremely fluent and flexible thinking, with creative content [new and original ideas], not necessarily centered on here and now experience".
Autobiographical Memory - The computerized version of the Autobiographical Memory Test (AMT; Williams et Broadbent, 1986). | The day before the beginning of the intervention
  This task focuses on retrieving past memories of personal events. A cue word appear on the computer screen. Participants have to click on a button as soon as they had retrieved a specific and autobiographical memory triggered by the cue word, in the time-limit of 1 minute after the cue onset. A window then appears to write the memory with as much specific and contextual details as possible. Before starting this task, participants are specified that the memory must have happened once and lasted less than 24 hours.After describing the memory, participants also have to judge (on a Likert type scale ranging from 0 to 10) the emotional intensity of the reported event. Moreover, they have to assess whether their memory was (1) pleasant, (2) unpleasant or (3) neutral. Finally, participants estimate the year during which this memory occurred.
  This AMT contains 6 French common nouns per time-measurement (3 success-relevant words, and 3 failure-relevant words) presented in a random order.
Autobiographical Memory - The computerized version of the Autobiographical Memory Test (AMT; Williams et Broadbent, 1986). | Once participants have completed 4 sessions of the intervention, about a week and a half after the beginning of the intervention
  This task focuses on retrieving past memories of personal events. A cue word appear on the computer screen. Participants have to click on a button as soon as they had retrieved a specific and autobiographical memory triggered by the cue word, in the time-limit of 1 minute after the cue onset. A window then appears to write the memory with as much specific and contextual details as possible. Before starting this task, participants are specified that the memory must have happened once and lasted less than 24 hours.After describing the memory, participants also have to judge (on a Likert type scale ranging from 0 to 10) the emotional intensity of the reported event. Moreover, they have to assess whether their memory was (1) pleasant, (2) unpleasant or (3) neutral. Finally, participants estimate the year during which this memory occurred.
  This AMT contains 6 French common nouns per time-measurement (3 success-relevant words, and 3 failure-relevant words) presented in a random order.
Autobiographical Memory - The computerized version of the Autobiographical Memory Test (AMT; Williams et Broadbent, 1986). | Two weeks after the end of the intervention
  This task focuses on retrieving past memories of personal events. A cue word appear on the computer screen. Participants have to click on a button as soon as they had retrieved a specific and autobiographical memory triggered by the cue word, in the time-limit of 1 minute after the cue onset. A window then appears to write the memory with as much specific and contextual details as possible. Before starting this task, participants are specified that the memory must have happened once and lasted less than 24 hours.After describing the memory, participants also have to judge (on a Likert type scale ranging from 0 to 10) the emotional intensity of the reported event. Moreover, they have to assess whether their memory was (1) pleasant, (2) unpleasant or (3) neutral. Finally, participants estimate the year during which this memory occurred.
  This AMT contains 6 French common nouns per time-measurement (3 success-relevant words, and 3 failure-relevant words) presented in a random order.
Autobiographical Memory - The computerized version of the Autobiographical Memory Test (AMT; Williams et Broadbent, 1986). | Three months after the end of the intervention
  This task focuses on retrieving past memories of personal events. A cue word appear on the computer screen. Participants have to click on a button as soon as they had retrieved a specific and autobiographical memory triggered by the cue word, in the time-limit of 1 minute after the cue onset. A window then appears to write the memory with as much specific and contextual details as possible. Before starting this task, participants are specified that the memory must have happened once and lasted less than 24 hours.After describing the memory, participants also have to judge (on a Likert type scale ranging from 0 to 10) the emotional intensity of the reported event. Moreover, they have to assess whether their memory was (1) pleasant, (2) unpleasant or (3) neutral. Finally, participants estimate the year during which this memory occurred.
  This AMT contains 6 French common nouns per time-measurement (3 success-relevant words, and 3 failure-relevant words) presented in a random order.
Multiple measures of Rumination state - State Repetitive Thoughts Questionnaire (SRTQ; Philippot et al., n.d.). | before the beginning of the intervention
  The SRTQ is a 10-item questionnaire, with a Likert type scale ranging from 1 ("totally disagree") to 5 ("totally agree"). It assesses the three modes of repetitive thinking (i.e., AERT, CERT, and CDRT) in their state form (i.e., subject to continuous changes and under many influences), in contrast with the RTMQ that assesses repetitive thinking as a stable individual characteristic.
Measure of change - Multiple measures of Rumination state - State Repetitive Thoughts Questionnaire (SRTQ; Philippot et al., n.d.). | Each day during the intervention, as well as between each week of the intervention
  The SRTQ is a 10-item questionnaire, with a Likert type scale ranging from 1 ("totally disagree") to 5 ("totally agree"). It assesses the three modes of repetitive thinking (i.e., AERT, CERT, and CDRT) in their state form (i.e., subject to continuous changes and under many influences), in contrast with the RTMQ that assesses repetitive thinking as a stable individual characteristic.
Measure of change - Multiple measures of Rumination state - State Repetitive Thoughts Questionnaire (SRTQ; Philippot et al., n.d.). | During two weeks after the end of the intervention, to assess the change from the 3-week intervention
  The SRTQ is a 10-item questionnaire, with a Likert type scale ranging from 1 ("totally disagree") to 5 ("totally agree"). It assesses the three modes of repetitive thinking (i.e., AERT, CERT, and CDRT) in their state form (i.e., subject to continuous changes and under many influences), in contrast with the RTMQ that assesses repetitive thinking as a stable individual characteristic.
Daily positive and negative emotions - Visual Analog Mood Scale (VAMS; McNally, Litz, Prassas, Shin, & Weathers, 1994). | before the beginning of the intervention.
  The VAMS is a seven-item questionnaire, with a Likert type scale ranging from 0 ("not at all") to 100 ("extremely"). It assesses the intensity of emotional states in the last few minutes: happy, sad, anxious, angry, emotionally aroused, in a positive mood, and in a negative mood. This questionnaire is used as a psychological distress measure.
Measure of change - Daily positive and negative emotions - Visual Analog Mood Scale (VAMS; McNally, Litz, Prassas, Shin, & Weathers, 1994). | Each day of the three-week intervention, to assess changes between the 10-day A-baseline phase and the intervention phase, as well as between each week of the intervention
  The VAMS is a seven-item questionnaire, with a Likert type scale ranging from 0 ("not at all") to 100 ("extremely"). It assesses the intensity of emotional states in the last few minutes: happy, sad, anxious, angry, emotionally aroused, in a positive mood, and in a negative mood. This questionnaire is used as a psychological distress measure.
Measure of change - Daily positive and negative emotions - Visual Analog Mood Scale (VAMS; McNally, Litz, Prassas, Shin, & Weathers, 1994). | During two weeks after the end of the intervention, to assess the change from the 3-week intervention
  The VAMS is a seven-item questionnaire, with a Likert type scale ranging from 0 ("not at all") to 100 ("extremely"). It assesses the intensity of emotional states in the last few minutes: happy, sad, anxious, angry, emotionally aroused, in a positive mood, and in a negative mood. This questionnaire is used as a psychological distress measure.

SECONDARY OUTCOMES:
Experiential avoidance - Multidimensional Experiential Avoidance Questionnaire (MEAQ ; Gamez, Chmielewski, Ruggero, Kotov, & Watson, 2011). | For the recruitment, i.e. until the number of 6 participants is reached for the second wave of the study (approximately two months after the beginning of the study)
  The MEAQ is a 62-items questionnaire with a Likert type scale ranging from 1 ("Totally disagree") to 6 ("Totally agree"). It assesses experiential avoidance with six different manifestations: Behavioral Avoidance (i.e., "overt, situational avoidance of physical discomfort and distress"), Distress Aversion (i.e., "negative evaluations or attitudes toward distress, nonacceptance of distress"), Procrastination (i.e., "delaying anticipated distress"), Distration/Supression (attempts to ignore or suppress distress"), Repression/Denial (i.e., "distancing and dissociating from distress, lack of distress awareness"), Distress Endurance (i.e., "willingness to behave effectively in the face of distress").
Experiential avoidance - Multidimensional Experiential Avoidance Questionnaire (MEAQ ; Gamez, Chmielewski, Ruggero, Kotov, & Watson, 2011). | The day before the beginning of the intervention
  The MEAQ is a 62-items questionnaire with a Likert type scale ranging from 1 ("Totally disagree") to 6 ("Totally agree"). It assesses experiential avoidance with six different manifestations: Behavioral Avoidance (i.e., "overt, situational avoidance of physical discomfort and distress"), Distress Aversion (i.e., "negative evaluations or attitudes toward distress, nonacceptance of distress"), Procrastination (i.e., "delaying anticipated distress"), Distration/Supression (attempts to ignore or suppress distress"), Repression/Denial (i.e., "distancing and dissociating from distress, lack of distress awareness"), Distress Endurance (i.e., "willingness to behave effectively in the face of distress").
Experiential avoidance - Multidimensional Experiential Avoidance Questionnaire (MEAQ ; Gamez, Chmielewski, Ruggero, Kotov, & Watson, 2011). | Once participants have completed 4 sessions of the intervention, about a week and a half after the beginning of the intervention
  The MEAQ is a 62-items questionnaire with a Likert type scale ranging from 1 ("Totally disagree") to 6 ("Totally agree"). It assesses experiential avoidance with six different manifestations: Behavioral Avoidance (i.e., "overt, situational avoidance of physical discomfort and distress"), Distress Aversion (i.e., "negative evaluations or attitudes toward distress, nonacceptance of distress"), Procrastination (i.e., "delaying anticipated distress"), Distration/Supression (attempts to ignore or suppress distress"), Repression/Denial (i.e., "distancing and dissociating from distress, lack of distress awareness"), Distress Endurance (i.e., "willingness to behave effectively in the face of distress").
Experiential avoidance - Multidimensional Experiential Avoidance Questionnaire (MEAQ ; Gamez, Chmielewski, Ruggero, Kotov, & Watson, 2011). | Two weeks after the end of the intervention
  The MEAQ is a 62-items questionnaire with a Likert type scale ranging from 1 ("Totally disagree") to 6 ("Totally agree"). It assesses experiential avoidance with six different manifestations: Behavioral Avoidance (i.e., "overt, situational avoidance of physical discomfort and distress"), Distress Aversion (i.e., "negative evaluations or attitudes toward distress, nonacceptance of distress"), Procrastination (i.e., "delaying anticipated distress"), Distration/Supression (attempts to ignore or suppress distress"), Repression/Denial (i.e., "distancing and dissociating from distress, lack of distress awareness"), Distress Endurance (i.e., "willingness to behave effectively in the face of distress").
Experiential avoidance - Multidimensional Experiential Avoidance Questionnaire (MEAQ ; Gamez, Chmielewski, Ruggero, Kotov, & Watson, 2011). | Three months after the end of the intervention
  The MEAQ is a 62-items questionnaire with a Likert type scale ranging from 1 ("Totally disagree") to 6 ("Totally agree"). It assesses experiential avoidance with six different manifestations: Behavioral Avoidance (i.e., "overt, situational avoidance of physical discomfort and distress"), Distress Aversion (i.e., "negative evaluations or attitudes toward distress, nonacceptance of distress"), Procrastination (i.e., "delaying anticipated distress"), Distration/Supression (attempts to ignore or suppress distress"), Repression/Denial (i.e., "distancing and dissociating from distress, lack of distress awareness"), Distress Endurance (i.e., "willingness to behave effectively in the face of distress").
Self-Discrepancy - Self-Discrepancies Scale (S-DS; Philippot, Dethier, Baeyens, & Bouvard, 2017). | For the recruitment, i.e. until the number of 6 participants is reached for the second wave of the study (approximately two months after the beginning of the study)
  The S-DS assesses the discrepancy between the perceived actual self (i.e., who people believe they are) and (a) the socially prescribe self (i.e., who people believe others would want them to be) or (b) the ideal self (i.e., who people ideally would want to be) (Philippot et al. 2017, p.3). Participants are first asked to write a maximum of 8 characteristics that they ideally wish to have (i.e., desired traits) and not have (i.e., undesired traits). They are provided a non-exhaustive sample of 105 characteristics, representing competence, likability, and physical appearance. Participants are then asked to estimate how much these characteristics currently define them (%). Finally, they are asked to indicate the extent to which the discrepancy between the perceived actual self and (a) the socially prescribe self or (b) the ideal self-generated distress, with a Likert type scale ranging to 0 ["I do not feel distress"] to 7 ["I feel significant distress"].
Self-Discrepancy - Self-Discrepancies Scale (S-DS; Philippot, Dethier, Baeyens, & Bouvard, 2017). | The day before the beginning of the intervention
  The S-DS assesses the discrepancy between the perceived actual self (i.e., who people believe they are) and (a) the socially prescribe self (i.e., who people believe others would want them to be) or (b) the ideal self (i.e., who people ideally would want to be) (Philippot et al. 2017, p.3). Participants are first asked to write a maximum of 8 characteristics that they ideally wish to have (i.e., desired traits) and not have (i.e., undesired traits). They are provided a non-exhaustive sample of 105 characteristics, representing competence, likability, and physical appearance. Participants are then asked to estimate how much these characteristics currently define them (%). Finally, they are asked to indicate the extent to which the discrepancy between the perceived actual self and (a) the socially prescribe self or (b) the ideal self-generated distress, with a Likert type scale ranging to 0 ["I do not feel distress"] to 7 ["I feel significant distress"].
Self-Discrepancy - Self-Discrepancies Scale (S-DS; Philippot, Dethier, Baeyens, & Bouvard, 2017). | Once participants have completed 4 sessions of the intervention, about a week and a half after the beginning of the intervention
  The S-DS assesses the discrepancy between the perceived actual self (i.e., who people believe they are) and (a) the socially prescribe self (i.e., who people believe others would want them to be) or (b) the ideal self (i.e., who people ideally would want to be) (Philippot et al. 2017, p.3). Participants are first asked to write a maximum of 8 characteristics that they ideally wish to have (i.e., desired traits) and not have (i.e., undesired traits). They are provided a non-exhaustive sample of 105 characteristics, representing competence, likability, and physical appearance. Participants are then asked to estimate how much these characteristics currently define them (%). Finally, they are asked to indicate the extent to which the discrepancy between the perceived actual self and (a) the socially prescribe self or (b) the ideal self-generated distress, with a Likert type scale ranging to 0 ["I do not feel distress"] to 7 ["I feel significant distress"].
Self-Discrepancy - Self-Discrepancies Scale (S-DS; Philippot, Dethier, Baeyens, & Bouvard, 2017). | Two weeks after the end of the intervention
  The S-DS assesses the discrepancy between the perceived actual self (i.e., who people believe they are) and (a) the socially prescribe self (i.e., who people believe others would want them to be) or (b) the ideal self (i.e., who people ideally would want to be) (Philippot et al. 2017, p.3). Participants are first asked to write a maximum of 8 characteristics that they ideally wish to have (i.e., desired traits) and not have (i.e., undesired traits). They are provided a non-exhaustive sample of 105 characteristics, representing competence, likability, and physical appearance. Participants are then asked to estimate how much these characteristics currently define them (%). Finally, they are asked to indicate the extent to which the discrepancy between the perceived actual self and (a) the socially prescribe self or (b) the ideal self-generated distress, with a Likert type scale ranging to 0 ["I do not feel distress"] to 7 ["I feel significant distress"].
Self-Discrepancy - Self-Discrepancies Scale (S-DS; Philippot, Dethier, Baeyens, & Bouvard, 2017). | Three months after the end of the intervention
  The S-DS assesses the discrepancy between the perceived actual self (i.e., who people believe they are) and (a) the socially prescribe self (i.e., who people believe others would want them to be) or (b) the ideal self (i.e., who people ideally would want to be) (Philippot et al. 2017, p.3). Participants are first asked to write a maximum of 8 characteristics that they ideally wish to have (i.e., desired traits) and not have (i.e., undesired traits). They are provided a non-exhaustive sample of 105 characteristics, representing competence, likability, and physical appearance. Participants are then asked to estimate how much these characteristics currently define them (%). Finally, they are asked to indicate the extent to which the discrepancy between the perceived actual self and (a) the socially prescribe self or (b) the ideal self-generated distress, with a Likert type scale ranging to 0 ["I do not feel distress"] to 7 ["I feel significant distress"].

OTHER OUTCOMES:
Intervention satisfaction - Consumer Satisfaction Questionnaire (QSC-8; Sabourin, Pérusse, & Gendreau, 1989). | Before each debriefing session with the experimenter
  The QSC-8 asseses how well the participant's needs regarding the intervention and its results are being met. It is an 8-item questionnaire with a Likert type scale ranging to 1 to 4, 4 being the maximum level of satisfaction.
Alcohol consumption - Alcohol Use Disorders Identification Test (AUDIT; Saunders, Aasland, Babor, DeLaFuente, & Grant, 1993) | The day before the beginning of the intervention
  The AUDIT is a 10-item screening questionnaire with an interval type scale of 3 or 4 choices. It assesses excessive drinking over the past week by focusing on three components: (a) alcohol intake, (b) alcohol dependence, and (c) alcohol-related problems.
Drug consumption - Drug Use Disorders Identification Test (DUDIT; Berman, Bergman, Palmstierna, and Schlyter, 2005). | The day before the beginning of the intervention
  The DUDIT is a 11-item screening questionnaire with an interval type scale of 3 or 4 choices. It assesses drug consumption over the past week to inform on two components: (a) drug intake, (b) symptoms criteria for substance abuse/harmful use and dependance according to the International Classification of Diseases (Tenth edition) and the Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition). A list of common illicit drugs as well as sedatives, hypnotics and analgesics is provided.
Daily drinking, cigarette use, and drug consumption - Timeline Followback (TLFB; Sobell & Sobell, 1992). | before the beginning of the intervention
  Participants first indicate whether they have used alcohol, cigarette, and/or drugs the day before and the day of the completion. If they answer "yes" for alcohol, cigarette, and / or cannabis they are then asked to specify quantities per day (i.e., number of alcohol glasses, and number of cigarettes or joints smoked). Participants are not required to quantify drugs due to (a) the lack of standardized assay units, (b) the wide range of purity and potency, as opposed to the percentage concentration requirement for alcohol products.
Measure of change - Daily drinking, cigarette use, and drug consumption - Timeline Followback (TLFB; Sobell & Sobell, 1992). | Each day of the three-week intervention, to assess changes between the 10-day A-baseline phase and the intervention phase, as well as between each week of the intervention
  Participants first indicate whether they have used alcohol, cigarette, and/or drugs the day before and the day of the completion. If they answer "yes" for alcohol, cigarette, and / or cannabis they are then asked to specify quantities per day (i.e., number of alcohol glasses, and number of cigarettes or joints smoked). Participants are not required to quantify drugs due to (a) the lack of standardized assay units, (b) the wide range of purity and potency, as opposed to the percentage concentration requirement for alcohol products.
Measure of change - Daily drinking, cigarette use, and drug consumption - Timeline Followback (TLFB; Sobell & Sobell, 1992). | During two weeks after the end of the intervention, to assess the change from the 3-week intervention
  Participants first indicate whether they have used alcohol, cigarette, and/or drugs the day before and the day of the completion. If they answer "yes" for alcohol, cigarette, and / or cannabis they are then asked to specify quantities per day (i.e., number of alcohol glasses, and number of cigarettes or joints smoked). Participants are not required to quantify drugs due to (a) the lack of standardized assay units, (b) the wide range of purity and potency, as opposed to the percentage concentration requirement for alcohol products.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Philippot, Principal Investigator — pierre.philippot@uclouvain.be
Locations (1):
- Université catholique de Louvain, Louvain-la-Neuve, Brabant Wallon, Belgium

IPD SHARING:
Plan to Share IPD: No
Data and analyses will be available from the investigators